CLINICAL TRIAL: NCT00495157
Title: Asthma Clinical Research Network (ACRN) Trial - Best Adjustment Strategy for Asthma in Long Term (BASALT)
Acronym: BASALT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Vernon M. Chinchilli, PhD, Professor and Chair, Department of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 494; 5U10HL074231 (NIH); U10HL074206 (NIH); U10HL074208 (NIH); U10HL074073 (NIH); U10HL074227 (NIH); U10HL074225 (NIH); U10HL074204 (NIH); U10HL074218 (NIH); U10HL074212 (NIH); U10HL074231 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Results first posted 2012-05-31 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Symptom-based adjustment (Experimental): Symptom-based adjustment of beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg or QVAR® 80 mcg)
  Interventions: Behavioral: Symptom-based adjustment
- Biomarker-based adjustment (Experimental): Biomarker-based adjustment of beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg or QVAR® 80 mcg)
  Interventions: Behavioral: Biomarker-based adjustment
- Guideline-based adjustment (Experimental): Guideline-based adjustment of beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg or QVAR® 80 mcg)
  Interventions: Behavioral: Guideline-based adjustment

INTERVENTIONS:
Behavioral: Symptom-based adjustment — Symptom-based adjustment of beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg or QVAR® 80 mcg)
  Arms: Symptom-based adjustment
Behavioral: Biomarker-based adjustment — Biomarker-based adjustment of beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg or QVAR® 80 mcg)
  Arms: Biomarker-based adjustment
Behavioral: Guideline-based adjustment — Guideline-based adjustment of beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg or QVAR® 80 mcg)
  Arms: Guideline-based adjustment

SUMMARY:
Asthma can be effectively controlled using inhaled corticosteroid medication. Treatment with inhaled corticosteroids often requires periodic adjustments to medication dosing and frequency levels. This study examines whether it is more beneficial to adjust corticosteroid treatment based on asthma symptoms and/or biomarkers of lung function versus standard medical guidelines.

DETAILED DESCRIPTION:
Asthma is a common, long-term disease that is caused by inflammation of the airways. Symptoms of asthma may include wheezing, coughing, shortness of breath, and chest tightness. The most common treatment for asthma is the use of inhaled corticosteroid medications with periodic adjustments to treatment intensity. For example, corticosteroid dosage is increased when asthma symptoms worsen and decreased when symptoms improve. However, guidelines for making these adjustments, especially reduced intensity adjustments, have not been well established. In people who are initially well controlled on daily low-dose inhaled corticosteroid therapy, symptom-based adjustment (SBA) and/or biomarker-based adjustment (BBA) of inhaled corticosteroid therapy may be more beneficial at maintaining asthma control than standard, guideline-based adjustments (GBA). The purpose of this study is to determine if adjusting treatment based on symptoms and/or lung function biomarkers is more effective at controlling asthma than adjusting corticosteroid use based on standardized medical guidelines.

This study begins with a 4-week period during which participants are monitored while they use an inhaler containing a low dose of inhaled corticosteroid medication. Participants then are assigned to take part in either the BASALT study or the Tiotropium as an Alternative to Long-Acting Beta-Agonists and Corticosteroids (TALC) study, which is a separate Asthma Clinical Research Network (ACRN) study. Participants in BASALT undergo 2 to 4 weeks of adherence testing, which involves using three inhalers that have electronic monitoring devices attached to them. Participants also are asked to measure and record their breathing rates and lung function in a study diary.

BASALT participants are then randomly assigned to one of three treatment groups: SBA, BBA, or GBA. Each participant is given four inhalers: one inhaler contains albuterol, which is used on an as-needed basis as rescue medication; one inhaler contains corticosteroid medication; and two inhalers contain placebo. One of the latter three inhalers is used each time the albuterol inhaler is used, and the other two inhalers are used on a daily basis. Study visits occur at Weeks 2, 4, 6, 12, 18, 24, 30, and 36 of the treatment period. Inhalers are adjusted during these visits based on SBA, BBA, or GBA guidelines. At selected visits, the following procedures occur: physical exam; blood collection; allergy skin testing; heart rate monitoring; lung function and airway testing; methacholine challenge test to determine asthma severity; and questionnaires to assess asthma control, quality of life, and other healthcare factors. Participants record asthma symptoms, peak flow measurements, and medication usage in a daily diary.

ELIGIBILITY:
Inclusion Criteria for BASALT and TALC Studies:

* Clinical history consistent with asthma
* Forced expiratory volume in one second (FEV1) greater than 40% of predicted value
* Asthma confirmed by one of the following two criteria:

  1. Beta-agonist reversibility to 4 puffs albuterol of at least 12% OR
  2. Methacholine provocative concentration at 20% (PC20) FEV1 of 8 milligrams per millimeter (mg/mL) or less when not on an inhaled corticosteroid, or 16 mg/mL or less when on an inhaled corticosteroid
* Need for daily controller therapy (i.e., inhaled corticosteroids, leukotriene modifiers, and/or long-acting beta-agonists) based on one or more of the following criteria:

  1. Received prescription for or used asthma controller within the 12 months prior to study entry OR
  2. Experienced symptoms for more than twice a week and not on asthma controller
* If on inhaled steroids (any drug at any dose not exceeding the equivalent of 1000 micrograms (mcg) of fluticasone daily), participant must have been on a stable dose for at least 2 weeks prior to study entry
* Non-smoker (i.e., total lifetime smoking history less than 10 pack-years; no smoking for at least 1 year prior to study entry)
* Willing to use an effective form of birth control throughout the study

Inclusion Criteria for BASALT Study:

* Ability to measure peak expiratory flow (PEF) each morning using the electronic peak flow meter (EPFM) device and to accurately transcribe the PEF measurements onto the diary cards at least 75% of the time during the last 2 weeks of the adherence testing period
* 75% compliance with recording peak flow measurements and symptoms in a symptom diary during the last 2 weeks of the adherence testing period
* Ability to take Inhalers A, B, and C at least 75% of scheduled doses; 75% compliance per inhaler is required
* No treatment failure (includes significant asthma exacerbation) within the last 4 weeks

Exclusion Criteria for BASALT and TALC Studies:

* Lung disease other than asthma, including chronic obstructive pulmonary disease (COPD) and chronic bronchitis
* Established or suspected diagnosis of vocal cord dysfunction
* Significant medical illness other than asthma
* History of respiratory tract infection within the 4 weeks prior to study entry
* History of a significant exacerbation of asthma within the 4 weeks prior to study entry
* History of life-threatening asthma requiring treatment with intubation and mechanical ventilation in the 5 years prior to study entry
* Hyposensitization therapy other than an established maintenance regimen
* Inability to coordinate use of the delivery devices used in the study, based on the opinion of the investigator or clinical coordinator
* Pregnant

Exclusion Criteria for BASALT Study:

* Inability to coordinate use of the medication delivery devices used in the study, based on the opinion of the investigator or clinical coordinator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2007-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Calhoun, MD, Principal Investigator — University of Texas, Galveston; Mario Castro, MD, Principal Investigator — Washington University School of Medicine; Robert F. Lemanske, MD, Principal Investigator — University of Wisconsin, Madison; Richard J. Martin, MD, Principal Investigator — National Jewish Health; Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital; Stephen P. Peters, MD, PhD, Principal Investigator — Wake Forest University Health Sciences; Homer A. Boushey, MD, Principal Investigator — University of California, San Francsico; Stephen I. Wasserman, MD, Principal Investigator — University of California, San Diego; Emily DiMango, MD, Principal Investigator — Columbia University; Monica Kraft, MD, Principal Investigator — Duke University; Reuben M. Cherniack, MD, Study Chair — National Jewish Health
Locations (10):
- United States (10):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Washington University, St. Louis, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - University of Wisconsin, Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Lugogo N, Green CL, Agada N, Zhang S, Meghdadpour S, Zhou R, Yang S, Anstrom KJ, Israel E, Martin R, Lemanske RF Jr, Boushey H, Lazarus SC, Wasserman SI, Castro M, Calhoun W, Peters SP, DiMango E, Chinchilli V, Kunselman S, King TS, Icitovic N, Kraft M. Obesity's effect on asthma extends to diagnostic criteria. J Allergy Clin Immunol. 2018 Mar;141(3):1096-1104. doi: 10.1016/j.jaci.2017.04.047. Epub 2017 Jun 15. PMID 28624608
- [Derived] Calhoun WJ, Ameredes BT, King TS, Icitovic N, Bleecker ER, Castro M, Cherniack RM, Chinchilli VM, Craig T, Denlinger L, DiMango EA, Engle LL, Fahy JV, Grant JA, Israel E, Jarjour N, Kazani SD, Kraft M, Kunselman SJ, Lazarus SC, Lemanske RF, Lugogo N, Martin RJ, Meyers DA, Moore WC, Pascual R, Peters SP, Ramsdell J, Sorkness CA, Sutherland ER, Szefler SJ, Wasserman SI, Walter MJ, Wechsler ME, Boushey HA; Asthma Clinical Research Network of the National Heart, Lung, and Blood Institute. Comparison of physician-, biomarker-, and symptom-based strategies for adjustment of inhaled corticosteroid therapy in adults with asthma: the BASALT randomized controlled trial. JAMA. 2012 Sep 12;308(10):987-97. doi: 10.1001/2012.jama.10893. PMID 22968888
- [Derived] Sutherland ER, Goleva E, Jackson LP, Stevens AD, Leung DY. Vitamin D levels, lung function, and steroid response in adult asthma. Am J Respir Crit Care Med. 2010 Apr 1;181(7):699-704. doi: 10.1164/rccm.200911-1710OC. Epub 2010 Jan 14. PMID 20075384
- See also: Click here for the Asthma Clinical Research Network Web site — http://www.acrn.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Symptom-based Adjustment | Biomarker-based Adjustment | Guideline-based Adjustment
Started | 113 | 115 | 114
Completed | 97 | 92 | 101
Not Completed | 16 | 23 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symptom-based Adjustment | Biomarker-based Adjustment | Guideline-based Adjustment | Total
Number analyzed (Participants) | 113 | 115 | 114 | 342
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 111 | 114 | 112 | 337
  >=65 years | 2 | 1 | 2 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 36.0 (12.2) | 34.8 (11.3) | 34.2 (11.9) | 35.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 82 | 72 | 237
  Male | 30 | 33 | 42 | 105
Region of Enrollment [Number; unit: participants]
  United States | 113 | 115 | 114 | 342

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure (Measured in Days)
Time Frame: Measured during the 36-week treatment period
Population: All participants were followed for time to treatment failure or right censoring (measured in days).
Measure: Mean (Standard Error); unit: days
Arm/Group | Symptom-based Adjustment | Biomarker-based Adjustment | Guideline-based Adjustment
Number analyzed (Participants) | 113 | 115 | 114
days | 196.9 (4.0) | 225.2 (5.6) | 182.3 (4.7)

2. Secondary Outcome: Number of Episodes of Treatment Failure
Time Frame: Measured during the 36-week treatment period
Reporting Status: Not Posted

3. Secondary Outcome: Time to First Asthma Exacerbation
Time Frame: Measured during the 36-week treatment period
Reporting Status: Not Posted

4. Secondary Outcome: Number of Asthma Exacerbations
Time Frame: Measured during the 36-week treatment period
Reporting Status: Not Posted

5. Secondary Outcome: Tests of Airway Caliber and Responsiveness (Forced Expiratory Volume in One Second (FEV1) Pre- and Post-bronchodilator Inhalation), Methacholine Provocative Concentration at 20% (PC20)
Time Frame: Measured during the 36-week treatment period
Reporting Status: Not Posted

6. Secondary Outcome: Tests of Airway Inflammation (Exhaled Breath Condensate (EBC), Fractional Exhaled Nitric Oxide (FeNO), Sputum Eosinophils)
Time Frame: Measured during the 36-week treatment period
Reporting Status: Not Posted

7. Secondary Outcome: Quality-of-life (AQLQ), Asthma Control Questionnaire (ACQ), and Number of Visit Days That ACQ is Less Than 1.25
Time Frame: Measured during the 36-week treatment period
Reporting Status: Not Posted

8. Secondary Outcome: Total Amount of Oral Prednisone Required and Total Amount of Inhaled Steroids
Time Frame: Measured during the 36-week treatment period
Reporting Status: Not Posted

9. Secondary Outcome: Adverse Events
Time Frame: Measured during the 36-week treatment period
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Symptom-based Adjustment | Biomarker-based Adjustment | Guideline-based Adjustment
Serious Adverse Events (participants affected / at risk) | 6/113 | 0/115 | 1/114
Other Adverse Events (participants affected / at risk) | 2/113 | 7/115 | 8/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symptom-based Adjustment (N=113) | Biomarker-based Adjustment (N=115) | Guideline-based Adjustment (N=114)
hospitalizations for unrelated events (General disorders) | 6 (6) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symptom-based Adjustment (N=113) | Biomarker-based Adjustment (N=115) | Guideline-based Adjustment (N=114)
urgent care for asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No